CLINICAL TRIAL: NCT07039539
Title: HARM REDUCTION PRACTICES AS AN INTERVENTION FOR PEOPLE USING ANABOLIC ANDROGENIC STEROIDS - THE RANDOMIZED CONTROLLED TRIAL NESTED INTO THE STUDY OF STEROIDS (SOS), THE PROSPECTIVE COHORT
Brief Title: HARM REDUCTION INTERVENTION FOR PEOPLE WHO USE ANABOLIC ANDROGENIC STEROIDS: THE RANDOMIZED CONTROLLED TRIAL
Acronym: SOS-RCT-HR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, President of the Center for Lifestyle Medicine - School of Medicine of University of São Paulo, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 77455824.7.0000.0068; 77455824.7.0000.0068 (Registry Identifier: SOS-RCT-HR)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Drug Abuse; Anabolic Steroids Adverse Reaction; Harm Reduction; Minimization, Harm
Keywords: human enhancement drug; performance and image enhancement drug; anabolic androgenic steroids; drug consumption; doping; harm reduction
MeSH Terms: conditions — Substance-Related Disorders; Harm Reduction

STUDY DESIGN:
Intervention Model Description: Intervention (harm reduction practices) and control (usual practices)
Who Masked: Outcomes Assessor
Masking Description: The researcher responsible for performing interviews will be blinded to the allocation of groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Harm Reduction intervention (Experimental): Will receive health care based on harm reduction paradigma
  Interventions: Behavioral: Harm Reduction intervention
- Control (No Intervention): Will receive regular and usual health care

INTERVENTIONS:
Behavioral: Harm Reduction intervention — Care intervention guided by the harm reduction paradigm. Based on the acceptance of participants' needs as a starting point for constructing care responses. Guidance will be provided in collective meetings with information based on reliable scientific evidence and will support the construction of new knowledge and practices of mutual support.
  Arms: Harm Reduction intervention

SUMMARY:
This study is about harm reduction (HR) practices for peolple who use anabolic androgenic steroids. It is a randomized controlled trial (RCT) that will compare a group that will receive an intervention in HR and another control (CTRL) that will receive usual guidelines. The primary outcome is the reduction in the final amount of drug consumed in relation to the initial planned amount. The secondary outcome is the understanding of what made the participants change their beliefs and change the planned pattern of AAS consumption.

DETAILED DESCRIPTION:
Introduction: This research is based on the analysis that the consumption of EAA has become a growing global concern due to the continuous increase in non-prescription consumption, illegalities and deaths. This can be noted by:

1. High global prevalence, approximately 3.3% of the global population has consumed or consumes EAA.
2. Significant increase in seizures by public security forces in the last year (2024-2025);
3. The circulation of information or misinformation on the subject in digital media, with special emphasis on social medias (Instagram and Facebook) and instant messaging groups (Telegram and Whatsapp); And the increase in outcomes of illness or even death related to the consumption of these drugs. This phenomenon seems to be on a rapid and worrying upward trend. On the other hand, it has been responded to slowly and with little effectiveness by actions such as, for example, "Bomba tô fora" (EAA, Im out), Bill Project 1236/2020, at the Brazilian federal level, which determines that gyms display signs, posters or banners about the harm caused by EAA, and even strictly prohibitive virtual games. As an institutional response, the Federal Council of Medicine published a clarification note 2333/2023, which contraindicated the use of EAA for aesthetic and physical performance purposes, under the justification that the abusive use of EAA increases the risk of cardiovascular accidents, sudden death and episodes of mental disorders. However, all of these initiatives are supported by sparse evidence and considered to be of low quality, with the most recent and robust evidence pointing to paths affiliated with HR, especially in the Netherlands, the United States, Norway and Australia. Therefore, taking on the task of constructing health responses to the phenomenon of EAA consumption in light of HR requires navigating moral debates that clash with the obvious ethical impossibility of prescribing such substances in supraphysiological doses to healthy humans. This is only possible with methodological rigor due to low-quality evidence, demanding multidimensional and combined work from various areas of health knowledge, but not only that, HR is also necessary.

This is the basis for this study 2, part of the consortium research: Abusive use of anabolic androgenic steroids in men and women: the SOS (Study of Steroid Abusers) cohort. SOS is a prospective cohort study with 200 participants to investigate the impacts of EAA consumption on general health in search of the best evidence for treatments, lines of care and prevention. Assuming that people have not stopped using AAS even with these contraindications and campaigns, then the imminent need for scientific production that answers, in the current reality, the questions present in this controlled intervention study is justified. Given the ethical limitations, we opted for a prospective cohort study with a broad approach carried out with habitual AAS users, that is, individuals who already plan or use AAS in their routine.

Then the question is: with which HR practices is the effectiveness of intervention confirmed for people who consume AAS? General objective: to investigate the effectiveness of the best HR-guided intervention practices for the consumption of AAS.

Specific objectives: to explore the phenomenon of AAS consumption in the health-disease process; to validate the HR instrument reporting resulting evidence to support the line of health care and public policies.

Experimental design: This is a randomized controlled trial (RCT) in which AAS consumers will undergo a HR intervention throughout their AAS use cycle. Participants will come from the prospective cohort study sample (SOS Study 1) and will be allocated to two groups, (i) intervention (HR) and (ii) control (CTRL). The primary outcome will be the reduction in AAS use, determined by the difference between the total dose of the cycle (in mg) planned at the beginning of the cycle (T0) and the dose actually consumed at the end (T1). As secondary outcomes, we will use qualitative methods to analyze the most effective practices based on the participants' perception. Data on changes in general health parameters identified in the battery of exams of the prospective cohort study (Study 1) will be used to compare the evaluation produced by the participants regarding the interventions.

Sample: When enrolled in the study, participants who plan to use for four weeks or longer will be informed in the informed consent form (ICF) about the possibility of being randomly allocated to the HR or CTRL groups to compose the sample of this RCT study. Those who occupy randomly distributed positions from position 50 to 100 may be included.

Thus, after the battery of health parameter assessments, at time T0 of the prospective cohort study, 36 participants will be allocated to either the HR (n = 18) or CTRL (n = 18) group. The sample size calculation was performed based on previous research with a design and objectives similar to those of the present study, but involving smokers (22), in which the effect size of the reduction in cigarette consumption was 1.6 (Cohen's d); assuming an alpha value of 0.05 and a power of 80%, 9 participants would be needed in each group. However, the sample in each group will be doubled to minimize the effect of possible dropouts throughout the study. The allocation of participants in each group will be randomized with the help of specific software (https://www.random.org/sequences/), in a 1:1 ratio, in blocks of four participants.

The inclusion criteria for AAS users are: no clinical indication for use, minimum age of 15 years, declared intention to use AAS for aesthetic or performance purposes within two weeks, and plan to use AAS for at least four consecutive weeks. The exclusion criterion is the use of AAS for sexual reassignment performed without clinical monitoring.

HR and CTRL intervention groups: The RD intervention will be carried out through six weekly meetings throughout the AAS cycle between the participants allocated to the HR group and the research team (23).

There will be an individual meeting before the start of the collective meetings. In these individual meetings, the first results of the HR group's health parameter tests can be discussed, any questions will be clarified and the participant will be encouraged to reflect about their EAA consumption, based on reliable scientific evidence. This is part of the perspective of action in HR and can be repeated as required by the participant allocated to the HR intervention group.

Then, the collective meetings of the HR intervention group will begin, which will be in the format of lectures given by health professionals, followed by discussion among the participants, in a circle. The topics covered will be self-organized based on the common demand for information among the participants. Additionally, the collective meetings may also address HR practices on related topics, for example: injection administration technique, substance testing and how to access reliable scientific information sources independently.

The six collective meetings will be planned to last an average of two hours in person, at FMUSP, in room 2223, second floor. In exceptional circumstances, a hybrid and synchronous format may be used (i.e., in-person for participants who can attend and remote for those who cannot). In cases of extreme need, such as the Covid-19 pandemic, meetings will be held entirely virtually, respecting the health requirements of restricting social contact.

The establishment of collective and individual meetings is based on the theoretical results of a previous study, in which EAA consumers were surveyed in order to understand the main points of an intervention for HR from the user's perspective. In this study, it was identified that HR actions should be focused on the user's health needs (24), such as:

(i) attention to one's own health; (ii) support network; (iii) pragmatic care strategies and; (iv) trust in health services. Attention to one's own health (i) will begin with health parameter tests, which will be explained in a humanized manner, ensuring full understanding of the content of the results. The support network (ii) will be formed by the interaction between participants and the research team in collective meetings. The care strategies (iii) will be designed by mediating the knowledge of the participants with the available scientific knowledge on the subject based on evidence.

The participants of the CTRL group, on the other hand, will take the assessment series during and after the EAA cycle and will receive all the information about the results and the risks associated with the use of EAA when receiving the results.

Participation in the CTRL group will not imply any omission of information or the necessary support from the team; only the approach will be affiliated with the usual care provided to this social group in the National Health System. After the end of the cycle, the data produced between HR and CTRL will be compared.

Outcomes: The primary outcome is the reduction in the use of AAS, which will be determined by the difference between the total dose of the cycle (in mg) that the participant planned to consume initially and the dose actually consumed at the end. As secondary outcomes, we will use qualitative indicators to analyze the practices. The most effective ones based on the participants' speech. The meetings will be recorded using audiovisual resources and, separately, the audio will be transcribed and submitted to a careful analysis to identify groups based on similarities.

The MAXQDA tool will be used to support content organization, triangulation, categorization, coding and analysis.

Adherence to the intervention would be also a important outcome because the more patient adheres to the conversation, accepts and understands what is being said, the more knowledge about the benefits and harms of AAS consumption can increase. This would contribute to greater knowledge, making them more discerning about their choices and positively impacting their overall quality of life.

Individual interviews: Individual interviews will be conducted with all participants in each group (HR and CTRL) before the start of the group meeting phase. Using the life story technique for the individual interview, it is possible to extract information and connections described by each participant in a more tailored manner to determine AAS consumption. This is because the life story seeks in the personal narrative an active reflection on the past, relating the individual experience and the social and historical context that determines the outcomes sought in this study.

After the experimental phase of the RCT (HR or CTRL), a new individual interview will be conducted in order to identify possible claims, concerns and questions about the approach tried (i.e. HR) or just monitoring (i.e. CTRL). The interviews will be in an open format, allowing free expression and chaining of the verbalized evaluation by the participant about what was experienced. The interviews will involve the participation of the researcher and the participant, and may take place either in person or remotely, according to the participant's availability. This is because it seems to be quite important that the individual interview after the experimental phase captures recent memories of the experience, avoiding loss of data or information that may be forgotten over time. The interviews will be recorded, with prior authorization from the participant, and transcribed for analysis.

Group meetings: Each HR or CTRL group, have a moderator and support team. The discussions will be recorded and transcribed for later qualitative analysis. The group activities will be in person, in a private room free from external noise, at FMUSP. The themes will be raised based on the discussion of the previous meeting, creating a link between one meeting and the next, to the same extent that it responds to exit needs constructed together with the participants.

Analysis of results: In both phases, content analysis will guide the process, which is defined as "a set of communication analysis techniques that aim to obtain, through systematic procedures and description of the content of the messages, indicators that allow inferring knowledge related to the conditions of production/reception of these messages". Initially, a cursory reading of the material will be carried out, followed by effective analysis with a deductive and inductive approach, characterizing two distinct forms of analysis, (i) classical and (ii) exploratory. Classical analysis is more deductive and uses categories (or themes) defined a priori and derived from theoretical frameworks. Exploratory content analysis will be characterized by a greater inductive aspect and the proposition that themes emerge from the data. The "cut and sort" approach will be used to identify themes, that is, a process that identifies important quotes and expressions and then organizes them into piles with similarities. Common factors will be identified, which will be used to formulate themes. Two researchers will independently carry out this entire process and reach a consensus on which themes were created/identified to build a repository of analytical categories.

MAXQDA software will be used to facilitate classical and exploratory analyses, both of individual interviews and group activities. For comparison between the two groups (i.e., RD and CTRL), panels will be constructed contrasting the themes.

ELIGIBILITY:
Inclusion Criteria:

* Anyone over 15 years of age
* Planning to use AAS for aesthetic or performance purposes
* Planned use for a period of four months or more

Exclusion Criteria:

* Use for medical indication for hypogonadism, for example
* Use for sexual reassignment

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Modulation of drug use | 2 months
  reduction in the total volume of drugs planned for the cycle compared to that used after the intervention (measured in milligrams of drugs)

SECONDARY OUTCOMES:
Decision-changing factors | 2 months
  Information declared by participants on motivations and changes in variables that led to changes in drug consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital of the School of Medicine, University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The results produced will be shared as requested by participants. All those who wish to be included will be included in a specific category in publications where this is possible.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the analysis is completed
Access Criteria: Having been a participant in the RCT